CLINICAL TRIAL: NCT01445119
Title: A Phase I Trial of Enzastaurin (LY317615) in Combination With Carboplatin in Adults With Recurrent Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 070053; 07-C-0053; NCT00438997 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Recurrent Gliomas
Keywords: Brain; Tumor; Radiation; Antiangiogenesis; Chemotherapy; Brain Tumor; Glioma
MeSH Terms: conditions — Glioma; Neoplasms; Brain Neoplasms | interventions — enzastaurin; Carboplatin

INTERVENTIONS:
Drug: Enzastaurin (LY317615)
Drug: Carboplatin

SUMMARY:
This study will evaluate the safety and effectiveness of Enzastaurin, an experimental drug that may prevent the growth of tumor vessels, in combination with Carboplatin, for patients who have a glioma, a type of brain tumor. Carboplatin is used for treating many kinds of cancers, though not recurrent gliomas. Tumor growth involves new cancer cell formation and accumulation, requiring a blood supply. Research shows that brain tumor cells can produce substances that stimulate new blood vessel formation. This study will look into whether the combination of drugs can stop that process.

Patients ages 18 and older who have recurring gliomas, who are not pregnant or breast feeding, and who do not have serious diseases may be eligible for this study. About 96 patients will participate for 1 year. They will have a physical examination, give blood and urine samples for analysis, and undergo magnetic resonance imaging (MRI) or computed tomography (CT) scans regarding tumor growth, and perhaps an electrocardiogram. Patients may also undergo a dynamic MRI with spectroscopy or PET scan (positron emission tomography), to distinguish a live tumor from a dying one. Researchers are studying patients taking a certain type of antiseizure medicine and patients who are not taking it because some antiseizure medicines may change the way the body handles a drug such as Enzastaurin. There will be two groups of participants, with 16 to 48 each. Group A is not taking enzyme-inducing antiseizure drugs, and Group B is taking such drugs. In Groups A and B are four dose levels, with 4 to12 patients at each level. Patients' doctors will tell them which group they belong to and how much Enzastaurin and Carboplatin they will take. Treatment consists of Enzastaurin every day for 5 weeks in Cycle 1 only and for 4 weeks beginning with Cycle 2 (each 4-week period as a cycle). Patients take Enzastaurin within 30 minutes after a meal. History, physical, and neurological examinations are repeated at the end of Cycle 1 and then every 4 weeks. Patients will have a repeat head MRI or CT scan before each cycle. If they tolerate the drugs without serious side effects and the tumor is not growing, they may continue with another cycle of Enzastaurin, taking the tablets every day, and Carboplatin being infused on Day 8 of Cycle 1 and on Day 1 of each additional cycle. Routine lab tests are done regularly. Patients will continue the 4-week cycles of treatment for as long as they have no serious side effects and there are no signs of tumor growth. Side effects of Enzastaurin may be fatigue, constipation, cough, and nausea. In men, there may be a decrease in sperm count. Carboplatin can lead to low counts in blood cells and platelets, and there may also be an allergic reaction. Vomiting is a likely side effect. At injection sites, there may be redness, swelling, and pain.

This study may or may not have a direct benefit for participants. However, information gained may help the sponsor of the study, Eli Lilly and Company, and may help patients in the future who have gliomas.

DETAILED DESCRIPTION:
Background:

* Enzastaurin, is a macrocyclic bisindolylmaleimide which disrupts the intrinsic phosphotransferase activity of conventional and novel PKC isoforms via an interaction at the ATP binding site, displays selectivity in inhibiting the isoforms. Preclinical studies demonstrate potent anti-angiogenic activity of enzastaurin and studies in normal volunteers and solid tumor patients demonstrate the drug is very well tolerated at doses that achieve a biologically active serum concentration.
* Carboplatin has shown activity as monotherapy in the treatment of recurrent malignant gliomas in adults and preclinical data generated in our laboratory demonstrates additive anti-glioma activity with enzastaurin. The safety profile of carboplatin and the preclinical and clinical data supports its use in combination with enzastaurin in patients with malignant gliomas.

Objective:

-To establish the maximally tolerated dose of enzastaurin in combination with carboplatin in patients with refractory primary brain tumors not on any enzyme-inducing anti-epileptic drugs (nEIAED) and for patients on EIAEDs.

Eligibility:

-Patients with histologically proven malignant glioma are eligible for this study.

Design:

-Patients will be stratified into two groups based on their anti-epileptic medications (nEIAEDs = Group A, EIAED = Group B)

Group A: Each cycle of therapy will consist of enzastaurin administered daily for 4 weeks with no breaks between cycles. All patients will receive a 7-day lead-in treatment period (Cycle 1) consisting of a loading dose of oral enzastaurin on Day 1 at 1125mg, followed by enzastaurin administered once daily at 500mg for 6 additional days in order to achieve steady state pharmacokinetics of enzastaurin. The first dose of carboplatin will be administered on Day 8 of Cycle 1, which will consist of 35 days. Following the lead-in treatment period, the first combination cycle of enzastaurin and carboplatin (Cycle 2) will commence as a 28-day cycle. Within each combination cycle, enzastaurin will be orally administered at 500mg once daily on Days 1 through 28 and carboplatin will be administered as an intravenous infusion over approximately 30 minutes on Day 1 every 28 days. The carboplatin dose will be 3 AUC for dose level one. For dose levels 2, 3, and 4, the carboplatin dose will be 4, 5 and 6 AUC, respectively.

Group B: Each cycle of therapy will consist of enzastaurin administered daily for 4 weeks with no breaks between cycles. All patients will receive a 7-day lead-in treatment period (Cycle 1) consisting of a loading dose of oral enzastaurin on Day 1 at 1125mg, followed by enzastaurin administered once daily at 875mg for 6 additional days in order to achieve steady state pharmacokinetics of enzastaurin. The first dose of carboplatin will be administered on Day 8 of Cycle 1, which will consist of 35 days. Following the lead-in treatment period, the first combination cycle of enzastaurin and carboplatin (Cycle 2) will commence as a 28-day cycle. Within each combination cycle, enzastaurin will be orally administered once daily on Days 1 through 28 at 875mg and carboplatin will be administered as an intravenous infusion over approximately 30 minutes on Day 1 every 28 days. The carboplatin dose will be 3 AUC for dose level one. For dose levels 2, 3, and 4, the carboplatin dose will be 4, 5 and 6 AUC, respectively.

National Cancer Institute (NCI) registered this trial with Eli Lilly as sponsor. NCI did not update the record. In June 2013, NCI transferred the trial to Lilly's clinicaltrials.gov account and Lilly updated the record with the trial status, study start date, and completion dates. This trial is not an applicable trial under Food and Drug Administration Amendments Act of 2007 (FDAAA).

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Patients with histologically proven malignant glioma who have progressive disease following standard treatment will be eligible for this protocol. Malignant glioma include glioblastoma multiforme (GBM), anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), anaplastic mixed oligoastrocytoma (AMO), or malignant glioma NOS (not otherwise specified). Additionally, patients with primitive neuroectodermal tumors (PNETs) of the central nervous system, progressive low-grade gliomas and radiographically diagnosed brain stem gliomas will be eligible.
2. Patients must have unequivocal evidence for tumor progression by MRI or CT scan. This scan should be performed within 14 days prior to registration and on a steroid dosage that has been stable for at least 5 days. If the steroid dose is increased between the date of imaging and registration a new baseline MR/CT is required. The same type of scan, that is., MRI or CT must be used throughout the period of protocol treatment for tumor measurement.
3. Patients having undergone recent resection of recurrent or progressive tumor will be eligible as long as all of the following conditions apply:

   A. They have recovered from the effects of surgery.

   B. Residual disease following resection of recurrent tumor is not mandated for eligibility into the study. To best assess the extent of residual disease post-operatively, a CT/ MRI should be done:
   * no later than 96 hours in the immediate post-operative period or
   * at least 4 weeks post-operatively, and
   * within 14 days of registration, and
   * on a steroid dosage that has been stable for at least 5 days.

   If the 96 hour scan is more than 14 days before registration, the scan needs to be repeated. If the steroid dose is increased between the date of imaging and registration, a new baseline MRI/CT is required on a stable steroid dosage for at least 5 days.
4. Patients must have failed prior radiation therapy and must have an interval of greater than or equal to 4 weeks from the completion of radiation therapy to study entry.
5. All patients or their previously designated LAR (Legally Authorized Representative) (if the patient is deemed by the treating physician to be cognitively impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) must sign an informed consent indicating that they are aware of the investigational nature of this study. Patients will be registered prior to starting the study.
6. Patients must be greater than or equal to 18 years old, and with a life expectancy greater than 8 weeks.
7. Patients must have a Karnofsky performance status of greater than or equal to 60.
8. Patients must have recovered from the toxic effects of prior therapy: 2 weeks from any noncytotoxic investigational agent, 4 weeks from prior cytotoxic therapy, two weeks from vincristine, 6 weeks from nitrosoureas, 3 weeks from procarbazine administration, and 1 week for non-cytotoxic agents, for example., interferon, tamoxifen, thalidomide, cis-retinoic acid, etc. (radiosensitizer does not count). Any questions related to the definition of non-cytotoxic agents should be directed to the Study Chair.
9. Patients must have adequate bone marrow function (WBC greater than or equal to 3,000/microl, ANC greater than or equal to 1,500/mm(3), platelet count of greater than or equal to 100,000/mm(3), and hemoglobin greater than or equal to 10 gm/dl), adequate liver function (SGOT and bilirubin less than or equal to 2 times ULN), and adequate renal function (creatinine less than or equal to 1.5 mg/dL and/or creatinine clearance greater than or equal to 60 cc/min) before starting therapy. These tests must be performed within 14 days prior to registration. Eligibility level for hemoglobin may be reached by transfusion.
10. Patients must not have any significant medical illnesses that in the investigator's opinion cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy.
11. This study was designed to include women and minorities, but was not designed to measure differences of intervention effects. Males and females will be recruited with no preference to gender. No exclusion to this study will be based on race.
12. Patients must practice adequate contraception.
13. Prior treatment with an enzyme inducing antiepileptic drug must have been discontinued at least 14 days prior to study entry for Group A patients.

EXCLUSION CRITERIA:

1. Patients who, in the view of the treating physician, have significant active cardiac, hepatic, or renal diseases are ineligible.
2. No concurrent use of other standard chemotherapeutics or investigative agents.
3. Prior treatment with platinum-based therapy.
4. Patients known to have an allergic response to mannitol.
5. Patients known to have an active malignancy other than their malignant glioma (except non-melanoma skin cancer or carcinoma in-situ of the cervix).
6. Patients who have an active infection requiring IV antibiotics.
7. Patients who are pregnant or breast feeding.
8. Patients who have any disease that will obscure toxicity or dangerously alter drug metabolism.
9. QTc with Bazett's correction that is unmeasurable, or greater than or equal to 460 msec on screening ECG. If a patient has QTc greater than or equal to 460 msec on screening ECG, a second screen ECG may be repeated at least 24 hours apart. The average QTc from the 2 screening ECGs must be less than 460 msec in order for the patient to be eligible for the study.
10. EKG demonstrating clinically significant arrythmia (multifocal premature ventricular contraction [PVC], bigeminy, trigeminy, ventricular tachycardia, bradycardia) that is symptomatic or requires treatment (CTCAE Grade 3), or asymptomatic sustained ventricular tachycardia.
11. Patients who have baseline EKGs suggestive of past or present cardiac ischemia will not be eligible unless they have an appropriate (as defined by the P.I. of this trial) negative cardiac work up (that is, echocardiogram, stress test).
12. Patients may not be on systemic anti-coagulants (that is, heparin, warfarin, small heparin fragments).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2007-01; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
To establish the maximally tolerated dose of enzastaurin in combination with carboplatin in patients with refractory primary brain tumors not on any enzyme-inducing anti-epileptic drugs (EIAED) and for patients on EIAEDs.

SECONDARY OUTCOMES:
To obtain exploratory data regarding the relationship between clinical outcome and GSK3-b activation in peripheral blood mononuclear cells in treated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Joohee Sul, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Soffietti R, Nobile M, Ruda R, Borgognone M, Costanza A, Laguzzi E, Mutani R. Second-line treatment with carboplatin for recurrent or progressive oligodendroglial tumors after PCV (procarbazine, lomustine, and vincristine) chemotherapy: a phase II study. Cancer. 2004 Feb 15;100(4):807-13. doi: 10.1002/cncr.20042. PMID 14770438
- [Background] Prados MD, Schold SC Jr, Fine HA, Jaeckle K, Hochberg F, Mechtler L, Fetell MR, Phuphanich S, Feun L, Janus TJ, Ford K, Graney W. A randomized, double-blind, placebo-controlled, phase 2 study of RMP-7 in combination with carboplatin administered intravenously for the treatment of recurrent malignant glioma. Neuro Oncol. 2003 Apr;5(2):96-103. doi: 10.1093/neuonc/5.2.96. PMID 12672281
- [Background] Prados MD, Warnick RE, Mack EE, Chandler KL, Rabbitt J, Page M, Malec M. Intravenous carboplatin for recurrent gliomas. A dose-escalating phase II trial. Am J Clin Oncol. 1996 Dec;19(6):609-12. doi: 10.1097/00000421-199612000-00016. PMID 8931682
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2007-C-0053.html